CLINICAL TRIAL: NCT06772688
Title: Evaluation of the Accuracy of Custom-made Plate in Maxillary Repositioning
Brief Title: Custom Made Plate in Orthognathic Surgery
Acronym: OGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Wafaa Anwar Mohamed Ali, Assistant lecturer, Faculty of Dental Medicine for Girls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OR SUR-108-2-N
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Maxillary Prognathism; Maxillary Retrusion
Keywords: Orthognathic surgery; Virtual planning; custom made plate
MeSH Terms: conditions — Retrognathia | interventions — Orthognathic Surgery

STUDY DESIGN:
Intervention Model Description: Fixation of maxilla with custom made plate designed by 3D virtual planning
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- designing of custom-made plate using 3Dvirtual planning (Experimental): patients underwent maxillary Le Fort I osteotomy using custom made plates for repositioning and fixation.
  Interventions: Procedure: orthognathic surgery

INTERVENTIONS:
Procedure: orthognathic surgery — Maxillary repositioning and fixation with custom made plate

SUMMARY:
Orthognathic surgery has traditionally been used to correct dentofacial deformities. Conventional methods rely on 2D radiographic images, occlusal splints, and dental casts, but these approaches have limitations, such as errors during face-bow transfer. Technological advancements, including 3D imaging, virtual surgical planning (VSP), and computer-aided design and manufacturing (CAD/CAM), have improved the precision and outcomes of orthognathic surgery.

DETAILED DESCRIPTION:
This study included one group of patients need orthognathic surgery and fixation of maxilla using custom made plate designed by 3D virtual planning using Materialize mimic soft ware

ELIGIBILITY:
Inclusion Criteria:

* Patients with skeletal class II or class III who need orthognathic surgery.
* Patients who suffer from clinical facial asymmetry.
* Patients with occlusal plane canting.
* Age range of patients 18-40 years old, with no gender prediction, able to read and sign the informed consent.

Exclusion Criteria:

* Maxillofacial trauma
* Patients who suffer from maxillofacial tumors
* Segmental maxillary surgery.
* Oral soft tissues defects, infections and bone metabolism disturbance.
* Allergy to titanium implant.
* Patient with systemic disease and immunocompromised patient.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the accuracy of custom-made plate | immediate postoperative
  CT to measure the accuracy

CONTACTS AND LOCATIONS:
Overall Officials: fatma ibrahim, Study Director — professor of oral and maxillofacial surgery
Locations (1):
- Faculty of dental medicine Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No